CLINICAL TRIAL: NCT00653822
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Single Dose Study to Assess the Tolerability, Safety, and Pharmacokinetics of Alefacept in Caucasian and Japanese Healthy Volunteers
Brief Title: A Study of Pharmacokinetics and Safety of Alefacept in Caucasian and Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 0485-CL-J101
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2008-08

CONDITIONS: Pharmacokinetics of Alefacept
Keywords: Amevive; alefacept; pharmacokinetics; Japanese
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1a (Experimental): IV
  Interventions: Drug: alefacept
- 1b (Placebo Comparator): IV
  Interventions: Drug: placebo
- 2a (Experimental): Lower SC dose
  Interventions: Drug: alefacept
- 2b (Placebo Comparator): SC to match lower dose
  Interventions: Drug: placebo
- 3a (Experimental): Higher SC dose
  Interventions: Drug: alefacept
- 3b (Placebo Comparator): SC to match higher dose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alefacept — IC and SC
  Other Names: Amevive; ASP0485
  Arms: 1a; 2a; 3a
Drug: placebo — IV and SC
  Arms: 1b; 2b; 3b

SUMMARY:
The objective of this study is to compare the pharmacokinetic and pharmacodynamic properties and safety profile of alefacept in Caucasian and Japanese healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or Japanese healthy subject with a body mass index (BMI) of 18 to 29 kg/m2, inclusive
* Japanese subject is first generation, born in Japan from parents of Japanese decent, and has resided outside of Japan for 5 years or less OR Caucasian subject is Hispanic or non-Hispanic, born of parents of European decent (not Mestizo or mixed race)
* Subject must have clinical laboratory test results within the normal therapeutic range or, if abnormal, the results are not clinically significant as determined by the investigator

Exclusion Criteria:

* CD4+ lymphocyte count outside normal limits at Screening
* Received vaccine within 60 days prior to study drug administration
* History of drug or alcohol abuse within the 2 years prior to the study drug administration
* Treatment with any systemic immunosuppressant agent within 6 months prior to study drug administration
* Treatment with any antibody or biologic product within 6 months prior to study drug administration
* Treatment with any systemic steroid or steroid inhaler within 2 months prior to study drug administration
* A smoking habit of greater than 10 cigarettes a day

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Serum alefacept pharmacokinetic parameters | Days 1-8,15, 22, 29 and 43

SECONDARY OUTCOMES:
Pharmacodynamic parameters of total lymphocyte count and peripheral lymphocyte subsets | Days 1-8, 15, 22, 29 and 43
Safety variables including anti-alefacept antibodies | Days 1-8, 15, 22, 29 and 43

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (1):
- Glendale, California, United States